CLINICAL TRIAL: NCT06388096
Title: CLAD Deconvolved PERG Responses in Glaucoma Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jorvec Corp. (Industry)
Collaborators: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: PERGCLAD001
Record Dates: First submitted 2024-04-22; First posted 2024-04-29 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Glaucoma, Suspect
Keywords: Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glaucoma Suspects (Experimental): Patients with suspicion of glaucoma based on positive factors of disease.
  Interventions: Diagnostic Test: Pattern Electroretinogram
- Controls (Active Comparator): Age matched controls to the glaucoma suspect group with no indications of glaucoma.
  Interventions: Diagnostic Test: Pattern Electroretinogram

INTERVENTIONS:
Diagnostic Test: Pattern Electroretinogram — Non-invasive recording of retinal potentials from a modulating pattern stimulus viewed on a visual display and recorded from surface electrodes around the eye.

SUMMARY:
Glaucoma is a progressive disease resulting in blindness. Determining the onset of the disease is critical so patients may obtain treatment to preserve useful vision. This study will collect data from a population of glaucoma suspects (with positive factors for the disease but with normal vision) along with a population of age matched controls using the pattern electroretinogram (PERG) and other standard eye tests for glaucoma. The PERG measures the function of retinal ganglion cells (RGCs) which come together to form the optic nerve. RGCs may become dysfunctional before dying. The Continuous loop deconvolution technique (CLAD) will be used to extract transient PERG responses in both glaucoma suspects and age matched controls. All patients will be monitored with PERG, Optic Coherence Tomography (OCT) and other ancillary tests over 2 years. CLAD will be compared with conventional techniques of monitoring glaucoma (standard PERG, OCT, visual field etc) to see if the CLAD is better at distinguishing between glaucoma suspects and controls.

DETAILED DESCRIPTION:
The PERG is recorded from small metallic cups taped on the skin or contact electrodes on the face similarly to an electrocardiogram except that the location is the skin around the eyes.

The only physical contact the subject will experience is a gentle cleaning of the skin with an alcohol prep pad. During the test the subject will be asked to look at a visual stimulus display for about 3 minutes. Depending on the experimental protocol, the subject may be asked to either sit during the test or to lie down in a bed. Lying down will cause a momentary increase of your eye pressure similar to the one that occurs during your normal sleep. This may help to understand whether or not your optic nerve functions normally when the pressure in your eye increases.

For OCT evaluation, the pupil will be dilated with drops similar to those used in a standard eye exam. The subject will have to briefly look at a mark inside the instrument one eye at a time.

For Visual field (VF) evaluation, the subject will be asked to look at a fixation mark inside the Visual Field testing equipment and asked to signal when they see small lights in their periphery.

PERG, OCT and VF will be performed during the same day of the visit. If the participant has already done these tests in the past, as part of another study or as part of standard treatment, the results of these tests will be obtained from shier record, and be included in this study.

RISKS:

For the PERG, the only significant risk to you is a small chance of skin discomfort from the cleansing agent for skin electrodes, which should go away without treatment. For OCT, there is a rare risk to you of an allergic reaction to the drops used to dilate your pupils. The risk is even lower if you did not have any reaction during your previous eye exams. In case of an allergic reaction, your eye doctor will immediately treat it. If you had previous problems with pupil dilation, you may wish to speak to your eye doctor about the option of doing this additional test. There are no significant risks associated with VF testing

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 85 years, inclusive
2. Refractive errors within -5 to +3 diopters
3. Best corrected visual acuity (BCVA) better than or equal to 20/30 (Snellen)
4. Normal standard automated perimetry (SAP) according to the Ocular Hypertension Treatment Study (OHTS) criteria15 (reliability < 15% on all indices, normality > 5% on all global indices in two consecutive sessions 6 months apart)
5. Minimum untreated Intraocular pressure IOP of 15 mm Hg
6. Glaucoma Suspect Status defined as one or more of the following:

   * Glaucomatous optic disc appearance (vertical cup-to-disc ratio [C/D] ≥0.5
   * Cup disc ratio asymmetry ≥0.2
   * Localized thinning of the disc
   * Presence or history of splinter disc hemorrhage
   * Moderately increased IOP (>21 to <28 mm Hg).
   * Family history of vision loss for glaucoma

Exclusion Criteria:

1. Age-related macular degeneration
2. Diabetes
3. Parkinson's disease
4. Multiple sclerosis
5. Unwilling or unable to give consent, unwilling to accept randomization, or unable to return for scheduled protocol visits.
6. Pregnant or nursing women.
7. Currently using prescribed pressure lowering medicines and unwilling to be withdrawn from them.
8. An OHTS risk score high enough in the judgment of the ophthalmologist or optometrist managing the patient to recommend pressure lowering medicine to the patient and not randomization.
9. An OCT abnormal enough in a pattern consistent with glaucoma.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
PERG Amplitude | Immediately after measurement
  Response amplitude measured in microvolts
PERG Latency | Immediately after measurement
  Response feature latency in milliseconds following the stimulus delivery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami, Bascom Palmer Eye Institute 900 NW 17th Street, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
The results from the project will be shared by presenting results at scientific conferences and publishing results in scientific journals. In addition, a de-identified database containing subject gender, age at recording, raw localization and tracking data, will be maintained. The data will be shared with other centers conducting similar research under appropriate IRB approval.
Supporting Information: Study Protocol
Time Frame: Data will be available six months after the completion of the project.

REFERENCES:
- [Background] Porciatti V, Feuer WJ, Monsalve P, Triolo G, Vazquez L, McSoley J, Ventura LM. Head-down Posture in Glaucoma Suspects Induces Changes in IOP, Systemic Pressure, and PERG That Predict Future Loss of Optic Nerve Tissue. J Glaucoma. 2017 May;26(5):459-465. doi: 10.1097/IJG.0000000000000648. PMID 28263259
- [Background] Porciatti V, Chou TH. Modeling Retinal Ganglion Cell Dysfunction in Optic Neuropathies. Cells. 2021 Jun 5;10(6):1398. doi: 10.3390/cells10061398. PMID 34198840
- [Background] Monsalve P, Ren S, Triolo G, Vazquez L, Henderson AD, Kostic M, Gordon P, Feuer WJ, Porciatti V. Steady-state PERG adaptation: a conspicuous component of response variability with clinical significance. Doc Ophthalmol. 2018 Jun;136(3):157-164. doi: 10.1007/s10633-018-9633-2. Epub 2018 May 19. PMID 29779071
- [Background] Monsalve P, Triolo G, Toft-Nielsen J, Bohorquez J, Henderson AD, Delgado R, Miskiel E, Ozdamar O, Feuer WJ, Porciatti V. Next Generation PERG Method: Expanding the Response Dynamic Range and Capturing Response Adaptation. Transl Vis Sci Technol. 2017 May 22;6(3):5. doi: 10.1167/tvst.6.3.5. eCollection 2017 May. PMID 28553559
- [Background] Toft-Nielsen J, Bohorquez J, Ozdamar O. Unwrapping of transient responses from high rate overlapping pattern electroretinograms by deconvolution. Clin Neurophysiol. 2014 Oct;125(10):2079-89. doi: 10.1016/j.clinph.2014.02.002. Epub 2014 Feb 14. PMID 24618216
- [Background] Ozdamar O, Toft-Nielsen J, Bohorquez J, Porciatti V. Relationship between transient and steady-state pattern electroretinograms: theoretical and experimental assessment. Invest Ophthalmol Vis Sci. 2014 Dec 4;55(12):8560-70. doi: 10.1167/iovs.14-15685. PMID 25477321